CLINICAL TRIAL: NCT06866028
Title: Enhancing Emotion Regulation Through fNIRS-informed Real-time Neurofeedback
Brief Title: Enhancing Emotion Regulation Through Functional Near-infrared Spectroscopy (fNIRS)-Informed Real-time Neurofeedback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HKU_NCAM_001
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Neurofeedback; Emotion Regulation; Stress
Keywords: fNIRS; emotion; neurofeedback
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Randomized sham-controlled parallel group fNIRS neurofeedback trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fNIRS neurofeedback training group (Experimental): Individuals in the fNIRS training group will receive feedback based on their real-time brain activity in the target region and learn to upregulate PFC activity while reappraising negative images.
  Interventions: Device: Real-time fNIRS neurofeedback from Turbo-Satori
- Sham training group (Sham Comparator): Individuals in the sham training group will receive yoked feedback from previous data acquired from another individual in real neurofeedback group while reappraising negative images.
  Interventions: Device: Yoked sham feedback from Turbo-Satori

INTERVENTIONS:
Device: Real-time fNIRS neurofeedback from Turbo-Satori — Activity in the target brain region measured by fNIRS in real-time will undergo processing on Turbo-Satori (BrainVoyager; Maastricht, Netherlands) to infer changes in oxygenated blood activity in the target brain region and relayed to the task program for visual feedback.
  Arms: fNIRS neurofeedback training group
Device: Yoked sham feedback from Turbo-Satori — Previous data acquired from another individual in the experimental group will be loaded into Turbo-Satori (BrainVoyager; Maastricht, Netherlands) software for preprocessing in real-time and relayed to the task program for visual feedback.
  Arms: Sham training group

SUMMARY:
The present study aims to employ real-time functional near-infrared spectroscopy (fNIRS) neurofeedback training in combination with cognitive reappraisal strategies for regulating negative emotions in healthy individuals.

Participants will complete:

* Cognitive reappraisal training with either real neurofeedback or sham feedback.
* Questionnaires at pre- and post- training timepoints
* A cold-pressor test at the end of the training

It is hypothesized that combining real-time fNIRS neurofeedback and cognitive reappraisal training will enhance emotion regulation in healthy individuals:

1. Increased neural activity in the prefrontal cortex (PFC) region of the brain will be significantly higher in the real neurofeedback group after training compared to the sham feedback group.
2. Real-time fNIRS-guided upregulation of the PFC will enhance emotion regulation during exposure to negative stimuli/scenes across the training runs.
3. The effects of fNIRS neurofeedback training will extend to influence emotion regulation in a cold-pressor test administered post-training, wherein individuals in the real neurofeedback group demonstrate better regulation of stress and pain induced by the task.

DETAILED DESCRIPTION:
The prevalence of stress-related disorders such as major depression and anxiety disorders has increased among children, adolescents and young adults internationally. Despite increasing concerns about the tremendous personal and societal toll of this development, efficacious interventions to reduce the detrimental impact of stress in young individuals are lacking. Therefore, working towards developing innovative approaches for regulating negative emotional experiences has substantial implications for addressing the prevailing mental health challenges affecting communities on a local and global scale.

Neurofeedback is a promising non-invasive neuromodulation technique allowing individuals to rapidly learn volitional control over brain activity via providing real-time feedback on brain function. Initial studies suggest that neurofeedback for emotion regulation produces increased experiences of positive emotion in patients with depression and decreased anxious mood in patients with anxiety disorder. A limitation of existing studies, however, is that neurofeedback training is often not directed with a concrete strategy that can help participants better learn control over brain activity, and extend learning outside of the experimental context.

Cognitive reappraisal, an emotion regulation strategy that focuses on reevaluating and changing the interpretation of an aversive scene or stimulus to reduce its negative impact on an individuals' emotions, has been implemented in several neurofeedback studies. It is shown to be effective in reducing negative emotions in clinical populations, such as in depression, anxiety, and trauma disorders when combined with fMRI neurofeedback. Meta-analytic evidence points to the lateral prefrontal cortex (lPFC) as a common region active during cognitive reappraisal. Thus, lPFC regions are a promising target for emotion regulation that has otherwise not been a target in existing studies, which traditionally focus on modulating emotional reactivity via subcortical regions.

Nevertheless, the implementation of neurofeedback-guided training on cortical level regions is relatively scarce, and even more so for improving emotion regulation in non-clinical populations. In our own previous studies, it has been previously demonstrated that healthy subjects can learn to control the activity of brain regions involved in emotional processing and that this can reduce anxiety. This suggests there is a promising potential of fNIRS neurofeedback training in combination with cognitive reappraisal strategies as a novel approach with broader implications for regulating stress in both clinical and non-clinical populations.

The present study aims to employ real-time fNIRS neurofeedback training in combination with cognitive reappraisal strategies for regulating negative emotions in healthy individuals. Participants will undergo cognitive reappraisal training with either real neurofeedback or sham feedback. Furthermore, emotion regulation ability will be assessed prior to and after neurofeedback training, through pre- and post-test behavioral measures and from comparing performance between real neurofeedback and sham feedback groups on a post-training task inducing physiological stress.

Participants will be explicitly instructed to apply cognitive reappraisal to upregulate brain activity. Prior to the neurofeedback runs, they will receive training illustrating the concept of cognitive reappraisal and neural basis of emotion regulation.

The present study will apply double-blinding. Participants will complete the experiment without knowing the presence of a control condition. The instructions administered to both groups will be exactly the same, and the experimenter responsible for administering instructions to the participant will not be aware of the participant's assigned group.

ELIGIBILITY:
Inclusion Criteria:

* Normal/corrected-to-normal vision
* Right-handed
* Below the cut-off for clinically-significant levels of depression (below 29) indicated by the Beck Depression Inventory (BDI-II; Beck et al., 1996)

Exclusion Criteria:

* Current/history of mental health conditions
* Current/history of chronic pain
* The following conditions: Cardiovascular disorder, Raynaud's phenomenon, fainting, seizure, wounds on the hand/arm
* Frequent use of alcohol/nicotine

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
Neurofeedback success on the neural level | 0 to 35 minutes following the start of the training
  Activity in the trained target brain region as measured by concomitant fNIRS (oxygenated signal) will be assessed over the four training runs, changes will be analyzed with analysis of variance (ANOVA) models.

SECONDARY OUTCOMES:
Effect on emotion regulation | 50-60 minutes following the start of the training
  Individuals will undergo an evaluated stress-induction procedure via the cold pressor test after the neurofeedback training. Effects on emotion regulation will be assessed using self-reported ratings of stress on visual analog scales ranging from 0-100 and analyzed using ANOVA models.
Effect on pain regulation | 50-60 minutes following the start of the training
  Individuals will undergo an evaluated stress-induction procedure via the cold pressor test after the neurofeedback training. Effects on pain regulation will be assessed using self-reported ratings of pain on visual analog scales ranging from 0-100 and analyzed using ANOVA models.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Jockey Club Building For Interdisciplinary Research, 5 Sassoon Rd, Sandy Bay, Hong Kong, Hong Kong

REFERENCES:
- [Background] Zweerings J, Sarkheil P, Keller M, Dyck M, Klasen M, Becker B, Gaebler AJ, Ibrahim CN, Turetsky BI, Zvyagintsev M, Flatten G, Mathiak K. Rt-fMRI neurofeedback-guided cognitive reappraisal training modulates amygdala responsivity in posttraumatic stress disorder. Neuroimage Clin. 2020;28:102483. doi: 10.1016/j.nicl.2020.102483. Epub 2020 Oct 28. PMID 33395974
- [Background] Zilverstand A, Sorger B, Sarkheil P, Goebel R. fMRI neurofeedback facilitates anxiety regulation in females with spider phobia. Front Behav Neurosci. 2015 Jun 8;9:148. doi: 10.3389/fnbeh.2015.00148. eCollection 2015. PMID 26106309
- [Background] Zilverstand A, Parvaz MA, Goldstein RZ. Neuroimaging cognitive reappraisal in clinical populations to define neural targets for enhancing emotion regulation. A systematic review. Neuroimage. 2017 May 1;151:105-116. doi: 10.1016/j.neuroimage.2016.06.009. Epub 2016 Jun 8. PMID 27288319
- [Background] Zhao Z, Yao S, Zweerings J, Zhou X, Zhou F, Kendrick KM, Chen H, Mathiak K, Becker B. Putamen volume predicts real-time fMRI neurofeedback learning success across paradigms and neurofeedback target regions. Hum Brain Mapp. 2021 Apr 15;42(6):1879-1887. doi: 10.1002/hbm.25336. Epub 2021 Jan 5. PMID 33400306
- [Background] Zhao Z, Yao S, Li K, Sindermann C, Zhou F, Zhao W, Li J, Luhrs M, Goebel R, Kendrick KM, Becker B. Real-Time Functional Connectivity-Informed Neurofeedback of Amygdala-Frontal Pathways Reduces Anxiety. Psychother Psychosom. 2019;88(1):5-15. doi: 10.1159/000496057. Epub 2019 Jan 30. PMID 30699438
- [Background] Yao S, Becker B, Geng Y, Zhao Z, Xu X, Zhao W, Ren P, Kendrick KM. Voluntary control of anterior insula and its functional connections is feedback-independent and increases pain empathy. Neuroimage. 2016 Apr 15;130:230-240. doi: 10.1016/j.neuroimage.2016.02.035. Epub 2016 Feb 17. PMID 26899786
- [Background] Pico-Perez M, Radua J, Steward T, Menchon JM, Soriano-Mas C. Emotion regulation in mood and anxiety disorders: A meta-analysis of fMRI cognitive reappraisal studies. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Oct 3;79(Pt B):96-104. doi: 10.1016/j.pnpbp.2017.06.001. Epub 2017 Jun 1. PMID 28579400
- [Background] COVID-19 Mental Disorders Collaborators. Global prevalence and burden of depressive and anxiety disorders in 204 countries and territories in 2020 due to the COVID-19 pandemic. Lancet. 2021 Nov 6;398(10312):1700-1712. doi: 10.1016/S0140-6736(21)02143-7. Epub 2021 Oct 8. PMID 34634250
- [Background] Linhartova P, Latalova A, Kosa B, Kasparek T, Schmahl C, Paret C. fMRI neurofeedback in emotion regulation: A literature review. Neuroimage. 2019 Jun;193:75-92. doi: 10.1016/j.neuroimage.2019.03.011. Epub 2019 Mar 9. PMID 30862532
- [Background] Keller M, Zweerings J, Klasen M, Zvyagintsev M, Iglesias J, Mendoza Quinones R, Mathiak K. fMRI Neurofeedback-Enhanced Cognitive Reappraisal Training in Depression: A Double-Blind Comparison of Left and Right vlPFC Regulation. Front Psychiatry. 2021 Aug 23;12:715898. doi: 10.3389/fpsyt.2021.715898. eCollection 2021. PMID 34497546
- [Background] Gross JJ. Emotion regulation: affective, cognitive, and social consequences. Psychophysiology. 2002 May;39(3):281-91. doi: 10.1017/s0048577201393198. PMID 12212647
- [Background] Buhle JT, Silvers JA, Wager TD, Lopez R, Onyemekwu C, Kober H, Weber J, Ochsner KN. Cognitive reappraisal of emotion: a meta-analysis of human neuroimaging studies. Cereb Cortex. 2014 Nov;24(11):2981-90. doi: 10.1093/cercor/bht154. Epub 2013 Jun 13. PMID 23765157